CLINICAL TRIAL: NCT05275686
Title: Effect of Novel Exhalational Delivery System With Fluticasone (EDS-FLU) on Eustachian Tube Dysfunction (ETD) in a Multi-center, Double-Blinded, Placebo-controlled Trial
Brief Title: Effect of Novel Exhalational Delivery System With Fluticasone (EDS-FLU) on Eustachian Tube Dysfunction (ETD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Sacramento Ear, Nose & Throat (Unknown); Ochsner Health System (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Arthur Wu, Principal Investigator, MD, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT-WU-2021-EuPEN
Record Dates: First submitted 2022-02-22; First posted 2022-03-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Eustachian Tube Dysfunction
Keywords: Eustachian Tube Dysfunction; Fluticasone
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Intervention Model Description: * Group 1 will get the EDS-FLU nasal spray and use at its normal twice a day dosing.
  * Group 2 will get the placebo nasal spray in an identical spray canister and use it twice a day.
  Patients will be randomized to receive placebo in the novel exhalation delivery system versus fluticasone in the device. Patients will take the spray twice daily for six weeks and then return for evaluation. An open label extension will be planned for both groups (placebo, non-placebo) at the end of the six weeks to use the EDS-FLU for an additional six weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and investigators will be kept blinded until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Placebo) (Placebo Comparator): Arm 1 (placebo) will get placebo spray per day.
  Interventions: Other: Placebo Nasal Spray
- Arm 2 (EDS-FLU) (Active Comparator): Arm 2 (EDS-FLU) will get 744 mcg of fluticasone propionate per day.
  Interventions: Drug: Fluticasone Propionate 93 MCG/1 ACTUATION Nasal Spray

INTERVENTIONS:
Drug: Fluticasone Propionate 93 MCG/1 ACTUATION Nasal Spray — Patients will use two sprays in each nostril twice a day for 6 weeks and additional 6 weeks (open label).
  Arms: Arm 2 (EDS-FLU)
Other: Placebo Nasal Spray — The Placebo is made of the following ingredients: Purified Water, Microcrystalline Cellulose RC-591, Dextrose, Anhydrous, EDTA Disodium Dihydrate, Benzalkonium Chloride Solution 50%, Polysorbate 80 (Tween 80, HP-LQ-(MH)), Sodium Hydroxide, and Hydrochloric Acid. Patients will use two sprays in each nostril twice a day
  Arms: Arm 1 (Placebo)

SUMMARY:
Intranasal nasal steroid sprays are the mainstay of treatment for chronic Eustachian tube dysfunction despite having little supportive evidence in the literature. A novel, commercially available nasal spray delivery system is available now for fluticasone that improves its delivery to the nasopharynx. The hypothesis of this study is that fluticasone using the novel spray system is effective for Eustachian tube dysfunction (ETD).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

Eustachian tube dysfunction (ETD) can be a symptom of allergic rhinitis, non-allergic rhinitis, or chronic rhinosinusitis. However, it can also be a separate entity with patients displaying no other symptoms of the previously mentioned diseases. There is currently no FDA- approved medication specifically for eustachian tube dysfunction, but most otolaryngologists, allergists, and primary care physicians employ multiple different over-the-counter and prescription medications for its treatment. Most common are oral and topical antihistamines, nasal steroid sprays, topical and oral decongestants, and oral steroids. Nasal steroid sprays, which are FDA-approved for allergic rhinitis, are most frequently used for chronic ETD despite a lack of large clinical trials to support their use. These sprays do have good safety profiles, are frequently available over-the-counter, and do have good data on their efficacy in rhinitis and sinusitis.

Fluticasone nasal spray is available over the counter and is a nasal steroid spray. It is frequently recommended or prescribed for chronic eustachian tube dysfunction. However, its efficacy and the efficacy of all nasal sprays may be limited by the access of previously available sprays into the nasopharynx. The level of evidence for these sprays in chronic ETD is poor overall with only one randomized controlled trial in adults. This study determined no benefit over placebo. In studies determining the deposition of nasal sprays, most of the spray is deposited in the front of the nasal cavity over the inferior turbinates and very little gets into the sinus cavities or nasopharynx. A new exhalational delivery system fluticasone spray (EDS-FLU) has been FDA-approved for patients with chronic rhinosinusitis with polyps. The main difference between this spray and previously available sprays is that it penetrates deeper into the sinuses and also to the nasopharynx, the location of the eustachian tubes. In this system, the user blows out while pumping the spray bottle and his/her breath is the driving force of the spray bottle. Blowing out also elevates the soft palate, seals the nasopharynx, and contains all the spray into the nasal cavity, sinuses, and nasopharynx. In a traditional spray, the soft palate is at resting position, and the spray can pass through the nasal cavity and down into the oropharynx and mouth. This is typically perceived by many users as postnasal drip after the use of nasal sprays. The investigators have previously published a retrospective review of the use of EDS-FLU in patients with at least 1 month of ETD symptoms and found that 79% had improvement more than the minimal clinically important difference. Thirty-six percent of patients normalized with regards to symptoms, and 80% of patients with pre- and post-treatment tympanometry normalized their tympanogram. This study will compare placebo to fluticasone exhalational nasal spray system (Xhance) in a randomized, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old, <80 years old
* Chronic Eustachian tube dysfunction defined as:

  * Symptoms in one or both ears > 3 months AND
  * ETDQ-7 score >14.5 AND
  * Type B, C, or As tympanometry
* Female subjects of childbearing potential must have a negative urine pregnancy test at screening and throughout the study duration.

Exclusion Criteria:

* Age <18 years old
* Known history of otologic surgery (excluding myringotomy or myringotomy tubes)
* Use of any additional intranasal medication
* Tympanic membrane perforation
* Adhesive otitis media
* Cholesteatoma or significant retraction pocket
* Middle ear effusion
* Nasopharyngeal tumor
* Any history of head and neck cancer
* Any history of head and neck irradiation
* Any history of temporomandibular disorder or prior surgery to the temporomandibular joint
* Any medical condition that the investigator deems inappropriate for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
7-Item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) | visit 2 (week 6)
  Eustachian tube dysfunction symptoms measured by the validated quality of life 7-Item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) at visit 2.
  The scale is from 1 (no problem) to 7 (severe problem).
7-Item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) | visit 3 (week 12)
  Eustachian tube dysfunction symptoms measured by the validated quality of life 7-Item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) at visit 3.
  The scale is from 1 (no problem) to 7 (severe problem).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Wu, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sacramento Ear, Nose & Throat, Sacramento, California
  - Indiana University, Indianapolis, Indiana
  - Ochsner Health System, New Orleans, Louisiana